CLINICAL TRIAL: NCT04223622
Title: Secretome from Mesenchymal Stem/stromal Cells on Human Osteochondral Explants: Cocktail of Factors Secreted by Adipose-derived Stromal Cells (ASC) for the Treatment of Osteoarthritis And/or for Articular Regeneration
Brief Title: Effects of ASC Secretome on Human Osteochondral Explants
Acronym: ASC-OA
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: ASC-OA
Record Dates: First submitted 2019-12-19; First posted 2020-01-10 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis
Keywords: mesenchymal stem/stromal cells; conditioned medium; extracellular vesicles; ASC
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: ASC secretome — The osteochondral explants isolated from arthroplasty patients will be induced to an OA phenotype and treated with ASC secretome (either complete conditioned medium or extracellular vesicles) in order to investigate its therapeutic potential.

SUMMARY:
Since the need of finding effective disease-modifying anti-osteoarthritis (OA) treatments is still unmet, with this study the investigators aim to gather further evidences of the therapeutic potential of Mesenchymal Stem/stromal Cell (MSC) secretome in order to pave the way to its future use as a cell-free biological product. In detail, the investigators predict to validate the promising results obtained in vitro, ex vivo on osteochondral explants, an OA model more representative of the physiological situation.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* age≥18 years old
* patients hospitalized in IRCCS (Istituto di Ricovero e Cura a Carattere Scientifico) Istituto Ortopedico Galeazzi, undergoing arthroplasty

Exclusion Criteria:

* age<18 years old
* patients unable to sign the Informed Consent
* positivity to serological test (HIV-Human Immunodeficiency Virus, HCV -Hepatitis C Virus, HBV -Hepatitis B Virus and TPHA -Treponema Pallidum Hemagglutination Assay)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Upon signing the Informed Consent, 24 male/female patients undergoing orthopedic surgery at IRCCS Istituto Ortopedico Galeazzi and matching the inclusion and esclusion criteria will be recruited.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Validation of the cell-free approach based on the use of ASC secretome on an ex vivo OA model by evaluation of cell viability, histological features and gene/protein expression of cartilage and bone biomarkers | 3 years
  Biochemical and functional characterization of untreated osteochondral explants (to set up the model) and explants treated with inflammatory cytokines (to simulate osteoarthritic pathology) by evaluation of several parameters. The multiple measurements that will concur to describe the phenotype of the specimens are the following:
  * cell viability by AlamarBlue (Arbitrary Fluorescence Units).
  * histological assessments (qualitative differences between specimens).
  * analysis of gene expression by RT-PCR (real-time polymerase chain reaction, relative quantification by 2-ΔΔCT method).
  * analysis of protein expression by Western Blot (relative quantification by densitometry) and Luminex (pg/ml).
  Evaluation of the effects of ASC secretome (either complete conditioned medium or its subcomponents) on osteochondral biopsies treated with inflammatory cytokines through the biochemical and functional analyses described above.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niada S, Giannasi C, Gomarasca M, Stanco D, Casati S, Brini AT. Adipose-derived stromal cell secretome reduces TNFalpha-induced hypertrophy and catabolic markers in primary human articular chondrocytes. Stem Cell Res. 2019 Jul;38:101463. doi: 10.1016/j.scr.2019.101463. Epub 2019 May 15. PMID 31108390
- [Derived] Cadelano F, Giannasi C, Rossi N, Della Morte E, Niada S, Talo G, Mistretta DA, Moretti M, Peretti GM, Mangiavini L, Brini AT, Choudhery MS. Evaluation of MSC-Secretome Effects in an Ex Vivo Compartmentalized Osteochondral Interface Model. Stem Cells Int. 2026 Jan 31;2026:3275855. doi: 10.1155/sci/3275855. eCollection 2026. PMID 41624062